CLINICAL TRIAL: NCT03609229
Title: Outcomes After Sacrocolpopexy With and Without Burch to Prevent Stress Urinary Incontinence in 3rd and 4th Degree Apical Uterine Prolapse. Randomized Controlled Trial
Brief Title: Outcomes After Sacrocolpopexy With and Without Burch to Prevent Stress Urinary Incontinence in 3rd and 4th Degree Apical Uterine Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCBU
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Prolapse
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Abdominal Sacrocolpopexy with burch technique
  Interventions: Procedure: Burch; Procedure: Abdominal Sacrocolpopexy
- control group (Active Comparator): Abdominal Sacrocolpopexy without burch technique
  Interventions: Procedure: Abdominal Sacrocolpopexy

INTERVENTIONS:
Procedure: Burch — polyglactin suture was passed through the Cooper's ligament bilaterally with the guidance of the valve
  Arms: Study group
Procedure: Abdominal Sacrocolpopexy — * By careful dissection (to avoid large veins in this region), expose the back of the pubic bone and the lateral aspects of the urethra.
  * The right-handed operator double gloves, and places the left hand in the vagina.
  * With fingers on either side of the catheter in the vagina, define the urethrovesical junction (at the balloon).
  * Place three Ethibond J-shaped sutures on either side of the urethrovesical junction.

SUMMARY:
Urinary incontinence will develop after prolapse repair in approximately one quarter of patients with advanced pelvic organ prolapse who remain continent despite significant loss of anterior vaginal and pelvic organ support. Many women with advanced pelvic organ prolapse who choose to undergo surgical management also choose to undergo continence surgery in order to prevent new onset urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

- Women with 3rd and 4th degree Apical prolapse

Exclusion Criteria:

* Patients with previous failed surgical intervention
* Patients with medical disorders that may interfere with surgical interventions .
* Patients with apical prolapsed complaining of stress urinary incontinence

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
the percentage of stress incontinence post operative | 3 months
  (symptoms, stress testing, or treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt